CLINICAL TRIAL: NCT02929901
Title: The Effects of Coffee Main Constituents (Caffeine and Chlorogenic Acid) Supplementation on Inflammatory, Metabolic Factors, Hepatic Steatosis and Fibrosis in None- Alcoholic Fatty Liver Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Dr Azita Hekmatdoost, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 147
Record Dates: First submitted 2016-10-09; First posted 2016-10-11 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Nonalcoholic Fatty Liver
MeSH Terms: interventions — Caffeine; Chlorogenic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- caffeine and chlorogeinc acid (Active Comparator): caffeine (200 mg) 1 capsule / day for 6 months plus chlorogenic acid (200 mg) 1 capsule / day for 6 months
  Interventions: Dietary Supplement: caffeine and chlorogenic acid
- caffeine (Active Comparator): caffeine (200 mg) 1 capsule / day for 6 months plus placebo (200) mg 1 capsule / day for 6 months
  Interventions: Dietary Supplement: caffeine
- chlorogenic acid (Active Comparator): chlorogenic acid (200 mg) 1 capsule / day for 6 months plus placebo (200 mg) 1 capsule / day for 6 months
  Interventions: Dietary Supplement: chlorogenic acid
- placebo (Placebo Comparator): placebo (200 mg) 1 capsule / day for 6 months plus placebo (200 mg) 1 capsule / day for 6 months
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: caffeine and chlorogenic acid — caffeine plus chlorogenic acid
  Arms: caffeine and chlorogeinc acid
Dietary Supplement: caffeine — caffeine plus placebo
  Arms: caffeine
Dietary Supplement: chlorogenic acid — chlorogenic acid plus placebo
  Arms: chlorogenic acid
Dietary Supplement: placebo — placebo plus placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the effects of coffee main constituents (caffeine and chlorogenic acid) supplements on inflammatory, metabolic factors, hepatic steatosis and fibrosis in none- alcoholic fatty liver patients with type 2 diabetes. Two hundred patients with fatty liver and type 2 diabetes will be randomly assigned to one of four groups: group 1, caffeine (200 mg/d) plus chlorogenic acid (200 mg/d); group 2, caffeine (200 mg/d) plus placebo; group 3, chlorogenic acid (200 mg/d) plus placebo; group 4, placebo plus placebo. Supplementation will be daily and will supervise for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with type 2 diabetes based on American Diabetes Association (ADA) definition or who only take oral antidiabetic drug.
* CAPscore >263

Exclusion Criteria:

* Criteria:

  * Taking any kind of antibiotics two weeks before recruitment;
  * History of alcohol consumption ;
  * pregnancy or lactation;
  * Professional athletes;
  * Other liver disease (viral/etc);
  * High dose synthetic estrogens, methotrexate , amiodarone, steroids, chloroquine, immunosuppressive drugs;
  * A history of Cardiovascular disease;
  * Renal disease, Celiac disease, Cirrhosis;
  * History of Upper Gastrointestinal surgery ;
  * A history of hypothyroidism or Cushing's syndrome;
  * History of drug dependence;
  * Body mass index (BMI) ≥35 kg/m2;
  * A restrictive diet or weight change ≥ 5 kg during the 3 months prior to study;
  * Any change in treatment with oral hypoglycemic; anti hypertensive and antilipid agents during the study;
  * Use of weight loss medications

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Hepatic steatosis | 6 months
  measured by CAP score using Fibroscan

SECONDARY OUTCOMES:
Glucose | 6 months
Glycated hemoglobin (HBA1C) | 6 months
alanine aminotransferase (ALT) | 6 months
aspartate aminotransferase (ALS) | 6 months
High sensitive C reactive protein ( hs- CRP) | 6 months
gut microbiota | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Iran

REFERENCES:
- [Derived] Mansour A, Mohajeri-Tehrani MR, Karimi S, Sanginabadi M, Poustchi H, Enayati S, Asgarbeik S, Nasrollahzadeh J, Hekmatdoost A. Short term effects of coffee components consumption on gut microbiota in patients with non-alcoholic fatty liver and diabetes: A pilot randomized placebo-controlled, clinical trial. EXCLI J. 2020 Mar 2;19:241-250. doi: 10.17179/excli2019-2021. eCollection 2020. PMID 32256270